CLINICAL TRIAL: NCT00484770
Title: Strategies for Tailoring Advanced Heart Failure Regimens in the Outpatient Setting: Brain Natriuretic Peptide Levels Versus the Clinical Congestion Score
Brief Title: STARBRITE: A Randomized Pilot Trial of BNP-Guided Therapy in Patients With Advanced Heart Failure
Acronym: STARBRITE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: American Heart Association (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4389; 0335132N
Record Dates: First submitted 2007-06-07; First posted 2007-06-11 (Estimated); Last update posted 2023-11-15 (Actual); Status verified 2007-06

CONDITIONS: Congestive Heart Failure
Keywords: heart failure, brain natriuretic peptide
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Congestion Score Strategy (Other)
  Interventions: Other: clinical assessment
- BNP Strategy (Other)
  Interventions: Device: Brain Natriuretic Peptide Levels -- Diagnostic testing; Other: clinical assessment

INTERVENTIONS:
Device: Brain Natriuretic Peptide Levels -- Diagnostic testing
  Arms: BNP Strategy
Other: clinical assessment

SUMMARY:
The primary hypothesis is that, in patients with advanced heart failure, an outpatient fluid management strategy guided by BNP levels and clinical targets will lead to fewer days hospitalized or dead over a 3-month period compared to an outpatient fluid management strategy using clinical targets alone.

DETAILED DESCRIPTION:
STARBRITE will test the hypothesis that a defined fluid management strategy, tailored to specific symptoms and physiological targets, will improve morbidity and mortality in the advanced heart failure population. Individual targets for each patient will be based on the outcome of the index hospitalization, during which therapy is adjusted to optimize clinical status, blood pressure, and renal function. Identifying a standard fluid management strategy may be an important way to limit the complications of diuretic therapy and the duration of hospitalization for these patients. In addition, a standard approach may provide objective criteria that can be used to systematically deliver care in many types of clinical settings.

In this study, patients will be randomized to two strategies of outpatient fluid management: 1) the Congestion Score Strategy and, 2) the BNP Strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted with NYHA class III/IV symptoms of heart failure
2. Left ventricular ejection fraction ≤35%
3. Will have received at least one dose of intravenous diuretics during the current hospitalization
4. Prior to discharge, has received heart failure education and has learned about daily weights, and fluid, sodium, and dietary restrictions
5. Able to return for follow-up care at the Brigham and Women's Hospital Cardiomyopathy Clinic or the Duke Heart Failure Management Program
6. Has regular access to a telephone
7. ≥18 years of age

Exclusion Criteria:

1. Moderate to severe valvular stenosis
2. Admitted with acute coronary syndrome
3. Creatinine >3.5
4. Renal failure on hemodialysis
5. Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2003-02; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Number of days neither hospitalized nor dead from the date of the first clinic visit to 90 days thereafter | 90 day follow up

SECONDARY OUTCOMES:
1. Number of days not dead from the date of the first clinic visit to 90 days thereafter 2.Number of days not hospitalized from the date of the first clinic visit to 90 days thereafter | 90 day follow up

CONTACTS AND LOCATIONS:
Overall Officials: Monica R Shah, MD, Principal Investigator — Duke University Medical Center/Washington Hospital Center

REFERENCES:
- [Result] Shah, MR for the STARBRITE Investigators. STARBRITE: A Randomized Pilot Trial of BNP-Guided Therapy in Patients with Advanced Heart Failure. Abstract. Circulation Supplement, October 2005. Presented at the American Heart Association Meeting in November 2005.